CLINICAL TRIAL: NCT01480999
Title: A Prospective Study Evaluating Surgical and Quality of Life Outcomes in Robotics and Laparoscopy Compared to Laparotomy in Early Stage Endometrial Cancer
Brief Title: Comparing Robotics and Laparoscopy With Laparotomy/Open Surgery for Endometrial Cancer
Acronym: GOC2
Status: Completed | Type: Observational
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Other Study IDs: 11-0447-CE
Record Dates: First submitted 2011-10-19; First posted 2011-11-29 (Estimated); Last update posted 2020-08-28 (Actual); Status verified 2020-08

CONDITIONS: Cancer of the Endometrium
Keywords: Laparotomy; Open Surgery; Laparoscopy; Robotic surgery
MeSH Terms: conditions — Endometrial Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- Laparotomy (open surgery)
- Laparoscopic surgery
- Robotic assisted surgery

SUMMARY:
The use of robotic surgery in the management of gynecologic cancers has increased exponentially in the United States since the implementation of technology in 2005. In Canada, access to the system is limited because of a lack of government funding. The government has been reluctant to fund this technology because robust data, on the true impact to patient care, is lacking.

This project will prospectively examine outcomes of women, with early stage endometrial cancer, treated surgically. Open surgery will be compared to minimally invasive surgery (MIS) which will include conventional laparoscopy and robotic surgery. The data collected will include detailed assessment of surgical data, peri-operative events, quality of life analysis, health economic evaluation and evaluation of MIS rates.

ELIGIBILITY:
Inclusion Criteria:

* Any type of histologically confirmed early stage (stage 1 or 2) cancer of the endometrium
* ECOG Performance status of 0-1
* Suitable candidate for surgery
* Signed approved informed consent
* Female, 18 years of age or older
* Pre-operative health is graded as ASA I-III
* Patients able to complete baseline questions either on their own or with assistance
* Patient willing to comply with scheduled visits

Exclusion Criteria:

* Major abdominal surgery, chemotherapy or radiation within 3 months before the baseline visit
* Evidence of diffuse peritoneal carcinomatosis by imaging or clinical exam
* Unfit for surgery: concomitant disorders incompatible with the study or surgery (at the discretion of the investigator)
* Patients who are breastfeeding or become pregnant during the study

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: New patients in the gynecologic oncology clinic will be offered the surgery that is deemed appropriate by their individual surgeon based on the patient's medical and surgical histories, type of malignancy, and the surgeon's expertise in open surgery, laparoscopy and/or robotic surgery.
Sampling Method: Non-Probability Sample
Enrollment: 550 (Actual)
Dates: Start 2011-11; Primary Completion 2015-07 (Actual); Study Completion 2020-08 (Actual)

PRIMARY OUTCOMES:
Surgical Outcomes | 6 months
  Intraoperative complications as well as perioperative (time to discharge from hospital), early postoperative (<4 weeks) and long-term morbidity (4 weeks to 6 months)
Quality of Life Outcomes | 6 months
  Validated quality of life questionnaires to assess the time it takes a patient to return to normal activity or work, the effect of surgery on their day-to-day living, pain, body image, sexuality, social life as well as about the costs associated with their surgery.
Cost-effectiveness | 6 months
  Compare cost-effectiveness between MIS (minimally invasive surgery) and open surgery for early stage endometrial cancer, by evaluating lengths of hospital stay, in hospital costs and out of hospital costs

SECONDARY OUTCOMES:
Evolution of MIS rates | Prior to recruitment of the first patient and every 6 months for the duration of the study
  Determine the evolution of MIS rates at each centre participating in this study, including the number of surgeons offering MIS, and the number of patients offered MIS. Evaluate whether the introduction of robotic surgery increases the proportion of patients undergoing MIS. Compare the characteristics of patients undergoing robotic-assisted, laparoscopic or open surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Marcus Q Bernardini, MD MSc FRCSC, Principal Investigator — Princess Margaret Hospital, University Health Network
Locations (7):
- Canada (7):
  - Cross Cancer Institute, Edmonton, Alberta
  - Kingston General Hospital, Kingston, Ontario
  - Sunnybrook Regional Cancer Centre, Toronto, Ontario
  - Princess Margaret Hospital, Toronto, Ontario
  - Hopital Notre-Dame du CHUM, Montreal, Quebec
  - Jewish General Hospital, Montreal, Quebec
  - Saskatoon Cancer Centre, Saskatoon, Saskatchewan